CLINICAL TRIAL: NCT03493412
Title: Effects of Tetrahydrobiopterin (BH4) on Leg Blood Flow, Mitochondrial Function and Leg Performance in Patients With Peripheral Artery Disease
Brief Title: Effects of Tetrahydrobiopterin (BH4) on Leg Blood Flow and Exercise Capacity in Patients With Peripheral Artery Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: discontinued due to change in operating plans prior to study initiation and enrollment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UNOmaha
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Artery Disease; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — sapropterin; Sugars

STUDY DESIGN:
Intervention Model Description: 1:1 Randomized, cross-over, double-blinded design
Who Masked: Participant, Investigator
Masking Description: Double-blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BH4-Placebo (Experimental): Subjects will be tested on two different days, first day will be baseline and Sapropterin Dihydrochloride (BH4, tetrahydrobiopterin) and second day will be Placebo. Testing will take place one-hour after BH4/placebo intake. There will be a 2-week washout between testing days.
  Interventions: Drug: Sapropterin Dihydrochloride (BH4, tetrahydrobiopterin); Drug: Placebo
- Placebo-BH4 (Experimental): Subjects will be tested on two different days, first day will be baseline and placebo and second day will be Sapropterin Dihydrochloride (BH4, tetrahydrobiopterin). Testing will take place one-hour after BH4/placebo intake. There will be a 2-week washout between testing days.
  Interventions: Drug: Sapropterin Dihydrochloride (BH4, tetrahydrobiopterin); Drug: Placebo

INTERVENTIONS:
Drug: Sapropterin Dihydrochloride (BH4, tetrahydrobiopterin) — 5 mg/kg will be used as the dose of BH4
  Other Names: 6R-BH4
Drug: Placebo — Placebo
  Other Names: Sugar Pill

SUMMARY:
Nitric oxide has been shown to be an important regulator within the cardiovascular system, responsible for regulation of blood flow, blood pressure and vascular growth. Cardiovascular diseases show a reduced ability of the peripheral blood vessels to dilate due to decreased levels of NO with concomitant increased levels of oxidative stress, which is extremely detrimental to patients with PAD, as the limited oxygen delivery to skeletal muscles ultimately results in claudication and reduced physical ability. However, this reduced oxygen delivery and utilization may be able to be improved as previous studies have revealed that tetrahydrobiopterin (BH4), is an important cofactor responsible for NO production. Furthermore, recent studies have shown that endothelial BH4 levels are associated with the vascular pathophysiological response to hypoxia, as it directly mediates endothelial nitric oxide synthase regulation and reduces superoxide production. Additionally, acute administration of BH4 was shown to improve vascular function, specifically, endothelial mediated vasodilatory function, in patients with systemic vascular and coronary disease, as well as six minute walking distances in patients with hypertension. Therefore, the purpose of this proposed study will be to examine the effects of BH4 on vascular function, oxidative stress and leg performance in patients with PAD. This study will examine patients with a classification of stage 1 or stage 2 peripheral artery disease who demonstrate a history of exercise-limiting claudication. Blood vessel oxygen transfer capacity in the leg will be assessed in the femoral and popliteal arteries with ultrasound, and blood vessel dilatory ability will be assessed in the brachial artery with flow-mediated dilation. Skeletal muscle mitochondrial function will be measured with near infrared spectroscopy, and ROS levels will be analyzed through blood samples. Leg function will be measured with an isokinetic dynamometer.

DETAILED DESCRIPTION:
According to the National Institute of Health, one in every twenty Americans over the age of 50 years old suffers from peripheral artery disease (PAD). PAD is a manifestation of systemic atherosclerosis and is specifically characterized by atherosclerotic blockages of the arteries in the legs. This results in claudication, a commonly experienced leg pain and immobility due to occlusion of the blood vessels. This pain reduces the amount of physical activity PAD patients can participate in, which can be detrimental to the patient, as it can lead to more systemic issues such as coronary artery disease, heart failure, and metabolic disorders, as well as amputation and death. These periods of occlusion are thought to be caused by endothelial dysfunction in the peripheral arteries leading to the legs, which results in an inability to produce nitric oxide (NO), a potent vasodilator which has been shown to be decreased in patients with PAD. Patients with PAD have also shown higher levels of systemic and skeletal muscle inflammation due to the impaired oxygen transfer capacity of these blood vessels. This inflammation leads to an increase in reactive oxygen species (ROS), which reduce the bioavailability of NO and are closely linked to the vascular dysfunction in PAD. Furthermore, mitochondria, a major cellular component that is responsible for the regulation between levels of production of ROS and antioxidants have shown to be altered in patients with PAD, which may lead to impaired oxygen transfer and utilization capacity, ultimately resulting in claudication, impaired functional capacity and reduced physical activity. Nitric oxide has been shown to be an important regulator within the cardiovascular system, responsible for regulation of blood flow, blood pressure and vascular growth. Additionally, many cardiovascular diseases have been shown to be highly associated with a reduced bioavailability of NO and a positively associated increase in ROS. These heightened levels of ROS not only reduce the availability of NO, but they may also cause cellular damage within the muscle and cardiovascular system. This combination of a reduced ability of the peripheral blood vessels to dilate due to decreased levels of NO, with a concomitant increased level of inflammation due to higher ROS levels could be extremely detrimental to patients with PAD, as the limited oxygen delivery to skeletal muscles could ultimately result in claudication and reduced physical ability. However, this reduced oxygen delivery and utilization may be able to be improved as previous studies have suggested that tetrahydrobiopterin (BH4), is an important cofactor responsible for NO production. Furthermore, recent studies have shown that endothelial BH4 levels are associated with the vascular pathophysiological response to hypoxia, as it directly mediates endothelial nitric oxide synthase regulation and reduces superoxide production. Additionally, acute administration of BH4 was shown to improve vascular function, specifically, endothelial mediated vasodilatory function, in patients with systemic vascular and coronary disease, as well as six minute walking distances in patients with hypertension. Therefore, the purpose of this proposed study will be to examine the effects of BH4 on vascular function, oxidative stress and leg performance in patients with PAD. The findings of this study may help to develop a new clinical therapy for patients with PAD. In this study we will examine endothelial function via flow-mediated dilation, blood flow in the femoral and popliteal arteries with a doppler ultrasound, leg skeletal muscle oxygenation with near-infrared spectroscopy, oxidative stress via blood samples and leg function by conducting a endurance test on an isokinetic dynamometer in 10 class-1 or class-2 PAD patients. We will use 5 mg/kg of BH4 obtained from Biomarin Pharmaceutical Industries in a 1:1 randomized, double-blinded, cross-over design with a 2-week washout period between testing days.

ELIGIBILITY:
Inclusion Criteria:

1. be able to give written, informed consent
2. demonstrate positive history of chronic claudication
3. have a history of exercise limiting claudication
4. have an ankle/brachial index < 0.90 at rest
5. have a stable blood pressure regimen, stable lipid regimen, stable diabetes regimen and risk factor control for 6 weeks.
6. be between 50-85 years old

Exclusion Criteria:

1. rest pain or tissue loss due to PAD (Fontaine stage III and IV)
2. acute lower extremity ischemic event secondary to thromboembolic disease or acute trauma
3. walking capacity limited by conditions other than claudication including leg (joint/musculoskeletal, neurologic) and systemic (heart, lung disease) pathology

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 2 days
  Flow-mediated dilation will be used to measure vasodilation in the brachial artery, and blood flow in the femoral and popliteal arteries

SECONDARY OUTCOMES:
Leg Function | 2 days
  Leg function will be measured with an isokinetic dynamometer
Oxidative Stress | 2 days
  Blood draws will be taken to measure oxidative stress markers in the blood
Skeletal Muscle Oxygenation | 2 days
  Near-infrared spectroscopy will be used to measure leg muscle oxygenation